CLINICAL TRIAL: NCT01121289
Title: A Trial Investigating the Pharmacokinetic Properties of NN1218 in Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating NN1218 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3808; U1111-1113-6955 (Other: WHO); 2009-017121-19 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- NN1218, formulation A (Experimental)
  Interventions: Drug: NN1218
- NN1218, formulation B (Experimental)
  Interventions: Drug: NN1218
- NN1218, formulation B (high) (Experimental)
  Interventions: Drug: NN1218
- NN1218, formulation C (Experimental)
  Interventions: Drug: NN1218
- NN1218, formulation D (Experimental)
  Interventions: Drug: NN1218
- insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: NN1218 — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: NN1218, formulation A
Drug: insulin aspart — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: insulin aspart
Drug: NN1218 — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: NN1218, formulation B
Drug: NN1218 — 0.4 U/kg body weight injected subcutaneously (under the skin)
  Arms: NN1218, formulation B (high)
Drug: NN1218 — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: NN1218, formulation C
Drug: NN1218 — 0.2 U/kg body weight injected subcutaneously (under the skin)
  Arms: NN1218, formulation D

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the absorption and effect in the body of NN1218 in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for more than 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for more than 12 months
* Body mass index (BMI) between 18.0-28.0 kg/m2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area under the serum NN1218 concentration-time curve | From 0-1 hours

SECONDARY OUTCOMES:
Area under the serum NN1218 concentration-time curve | From 0-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com